CLINICAL TRIAL: NCT05371535
Title: A Prospective, Randomized, Multi-center, Parallel Controlled Trial Evaluating the Efficacy and Safety of MatrixOssTM Bone Graft in Bone Defect Repair Caused by Tooth Extraction
Brief Title: A Clinical Trial to Evaluate the Safety and Effectiveness of MatrixOssTM Bone Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Collagen Matrix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WCHSIRB-D-2022-154
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Dental Diseases
MeSH Terms: conditions — Stomatognathic Diseases

STUDY DESIGN:
Intervention Model Description: Subjects included will be randomly assigned into the experimental group and the control group at a ratio of 1:1. Those in the experimental group will receive MatrixOssTM Bone Graft plus Bio-Gide membrane, and those in the control group will receive Bio-Oss Bone Graft plus Bio-Gide membrane.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Experimental group (Experimental): Those in the experimental group will receive MatrixOssTM Bone Graft plus Bio-Gide membrane.
  Interventions: Device: MatrixOssTM Bone Graft plus Bio-Gide membrane
- Control group (Active Comparator): Those in the control group will receive Bio-Oss Bone Graft plus Bio-Gide membrane
  Interventions: Device: MatrixOssTM Bone Graft plus Bio-Gide membrane

INTERVENTIONS:
Device: MatrixOssTM Bone Graft plus Bio-Gide membrane — To verify the efficacy and safety of MatrixOssTM Bone Graft developed and manufactured by Collagen Matrix, Inc. for bone defect repair caused by tooth extraction.

SUMMARY:
The objective of this clinical trial is to evaluate the efficacy and safety of MatrixOssTM Bone Graft in bone defect repair caused by tooth extraction.

DETAILED DESCRIPTION:
This is a prospective, randomized, multi-center and parallel controlled clinical trial. It is planned to be carried out in more than 3 (including 3) hospitals with qualifications as a national-level clinical trial institution. Subjects included will be randomly assigned into the experimental group and the control group at a ratio of 1:1. Those in the experimental group will receive MatrixOssTM Bone Graft plus Bio-Gide membrane, and those in the control group will receive Bio-Oss Bone Graft plus Bio-Gide membrane. To evaluate whether the changes in alveolar ridge height from baseline to 24 weeks postoperative in the experimental group is non-inferior to that in the control group, so as to verify the efficacy and safety of MatrixOssTM Bone Graft developed and manufactured by Collagen Matrix, Inc. for bone defect repair caused by tooth extraction.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18-65 years (including 18 years and 65 years);
2. Bone loss caused by singe tooth extraction requiring bone grafting;
3. At least one natural tooth adjacent to the targeted tooth;
4. The subjects could understand the purpose of this trial, voluntarily participate in this trial and willing to sign an Informed Consent Form (ICF).

Exclusion Criteria:

1. Bone defect caused by invasive or malignant bone tumors；
2. Subjects with uncontrolled periodontitis, acute periapical inflammation;
3. Subjects who are receiving or had received any drug in last 3 months that may influence or promote bone metabolism;
4. Active infectious disease, various bone defects during the active phase of metabolic bone disease;
5. Subjects with acute or chronic infection (osteomyelitis) at the surgical site;
6. Subjects with osteoporosis or osteomalacia;
7. Alanine Aminotransferase，ALT）Aspartate Aminotransferase，AST） Subjects with abnormal liver or kidney functions (ALT or AST or creatinine exceeds 1.5 times the upper limit of normal range);
8. Subjects who has a history of or is undergoing cervico-facial radiotherapy or chemotherapy;
9. Subjects with serious blood system diseases, such as leukemia or other hemorrhagic diseases;
10. Subjects with abnormal coagulation function;
11. Subjects with severe cardiovascular and cerebrovascular diseases;
12. Subjects with systemic diseases may affect postoperative healing and/or osseointegration, such as diabetes, uncontrolled hypertension (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg), hyperparathyroidism, etc.
13. Subjects with mental disorder and lack of behavioral autonomy;
14. Known allergy or hypersensitivity to animal-derived implantable materials;
15. Subjects who refuse to use porcine-derived implantable materials;
16. Pregnant and lactating women, or those who plan to conceive within 6 months;
17. Subjects with implants adjacent to the targeted teeth that can cause oral imaging artifacts, such as metal dentures, porcelain teeth, etc. that may cause oral imaging artifacts;
18. Subjects who smoking more than 5 cigarettes per day;
19. Subjects who are alcoholism, drug abuse, or drug dependence;
20. Subjects who have participated or are participating in a drug clinical trials in last 3 months, or have participated in other medical device clinical trials in last 30 days;
21. Other circumstances which are considered by the investigator not suitable for enrollment in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2022-05-30 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in alveolar ridge height from baseline to 24 weeks postoperative. | 24 weeks
  The alveolar ridge height immediately postoperative and 24 weeks postoperative were measured by CBCT, and changes in alveolar ridge height were calculated. Evaluate whether the changes in alveolar ridge height 24 weeks postoperative in the experimental group was non-inferior to that in the control group.

SECONDARY OUTCOMES:
Changes in alveolar ridge width from baseline to 24 weeks postoperative | 24 weeks
  The alveolar ridge height immediately postoperative and 24 weeks postoperative were measured by CBCT, and changes in alveolar ridge height were calculated. Compare the changes in alveolar ridge width from baseline to 24 weeks postoperative between the experimental group and control group.
Bone graft density in alveolar socket 24 weeks postoperative | 24 weeks
  According to the CBCT results at 24 weeks postoperative, the consistency between the bone graft density in alveolar socket and the surrounding alveolar bone density was evaluated. The evaluation contents include:
  1. Lower than surrounding alveolar bone density;
  2. Same as surrounding alveolar bone density;
  3. Higher than surrounding alveolar bone density.
Wound healing | 10 days postoperative and 4 weeks postoperative
  The wound healing conditions of the subjects in the experimental group and control group 10 days postoperative and 4 weeks postoperative were assessed using the Wound Healing Assessment Scale, and the gingival tissue in the implanted area of the material was evaluated as follows:
  Score 1 = uneventful healing with no gingival edema, erythema, suppuration, patient discomfort, or flap dehiscence; Score 2 = uneventful healing with slight gingival edema, erythema, patient discomfort, or flap dehiscence but no suppuration; Score 3 = poor wound healing with significant gingival edema, erythema, patient discomfort, flap dehiscence, or any suppuration.
Rejection reaction | 12 weeks
  Observe whether there are redness, suppuration, inflammation, granulation tissue hyperplasia, exposure/overflow of bone graft and other rejection reactions at the operation site of the subjects in the experimental group and the control group from immediately to 12 weeks postoperative.
Device performance evaluation | 24weeks
  The device performance of the experimental device/control device was evaluated by the investigator, and the evaluation criteria were as follows:
  Is the product operation convenient?
  * Convenient
  * Common
  * Inconvenient
    （2）Is the product easy to fuse with blood?
  * Easy to fuse
  * Common
  * Not easy to fuse

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jian Pan, Principal Investigator — West China Stomatological Hospital of Sichuan University

IPD SHARING:
Plan to Share IPD: No